CLINICAL TRIAL: NCT02986165
Title: Efficacy of a Tomato Pomace Extract for Inhibiting Platelet Aggregation
Brief Title: Effect of Ingesting a Tomato Pomace Extract on Platelet Aggregation
Acronym: Tomasa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Estudios en Alimentos Procesados (Other)
Collaborators: University of Talca (Other); Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R15F10012
Record Dates: First submitted 2016-11-23; First posted 2016-12-08 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Diseases
Keywords: Platelet Aggregation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo control (Placebo Comparator): 100 g of flavoured water
  Interventions: Dietary Supplement: Placebo control
- Low dose pomace extract (Experimental): 1 g pomace extract powder
  Interventions: Dietary Supplement: Low dose pomace extract
- High dose pomace extract (Experimental): 2.5 g pomace extract powder
  Interventions: Dietary Supplement: High dose pomace extract

INTERVENTIONS:
Dietary Supplement: Placebo control — The placebo control is water containing a commercially available orange flavoured powder (Kool aid) which will be diluted according to the manufacturer's instructions
  Arms: Placebo control
Dietary Supplement: Low dose pomace extract — Immediately prior to ingestion, 'drinks' containing 1 g of tomato pomace extract will be prepared at the research facility. The water used to dilute the extract will be flavoured using a commercially available orange flavoured powder (Kool aid) which will be diluted according to the manufacturer's instructions before adding to the tomato pomace extract.
  Arms: Low dose pomace extract
Dietary Supplement: High dose pomace extract — Immediately prior to ingestion, 'drinks' containing 2.5 g of tomato pomace extract will be prepared at the research facility. The water used to dilute the extract will be flavoured using a commercially available orange flavoured powder (Kool aid) which will be diluted according to the manufacturer's instructions before adding to the tomato pomace extract.
  Arms: High dose pomace extract

SUMMARY:
This study evaluates the acute and longer term effects of a tomato pomace extract on platelet aggregation in health subjects.

DETAILED DESCRIPTION:
Evidence from human intervention trials and mechanistic studies suggests that tomato and tomato based products are associated with a reduction in CVD risk. The mechanism by which this protective effect occurs is not clearly understood but research has focused on its potential to modulate platelet function. This single-blind, randomized, parallel design human intervention trial will recruit 99 participants to consume an orange flavoured beverage containing different doses of a tomato pomace extract (1.0 and 2.5 g) or placebo control over a 5-day period. The study aims is to investigate the effects of consuming different doses of the tomato pomace extract on platelet aggregation. Safety and tolerability of the tomato pomace extracts was tested prior starting this study by undertaking a single ascending dose study.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men aged between 18 and 26 years
* BMI >19.5 and <26.0
* Platelet aggregation response corresponding to ≥ 65%

Exclusion Criteria:

* Known tomato allergy
* Chronic medical conditions requiring active treatment (e.g. cardiovascular disease, diabetes, asthma)
* Gastro-intestinal disease/disorders
* Smokers
* Medically prescribed medication known to affect platelet function
* Self-prescribed medication known to affect platelet function (e.g. aspirin and non-steroidal anti-inflammatory drugs) unless participant is willing to give up.
* Bleeding disorders (e.g. haemophilia)
* Dietary supplements judged to affect study outcome
* Parallel participation in another research project which involves dietary intervention
* Blood donation within 16 weeks prior to the study
* Depressed or elevated blood pressure measurements (<90/50 or 95/50 if symptomatic or ≥ 160/100 mmHg)
* Any person related to or living with any member of the study team

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline platelet aggregation at three hours | Blood samples on two separate occasions (baseline and three hours post-intervention)

SECONDARY OUTCOMES:
Change from baseline platelet aggregation at 5 days | Blood samples on two separate occasions (baseline and 5 days post- intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Palomo, Dr., Principal Investigator — University of Talca
Locations (1):
- University of Talca, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law MR, Morris JK. By how much does fruit and vegetable consumption reduce the risk of ischaemic heart disease: response to commentary. Eur J Clin Nutr. 1999 Nov;53(11):903-4. doi: 10.1038/sj.ejcn.1600944. PMID 10557006
- [Background] Ruggeri ZM. Platelets in atherothrombosis. Nat Med. 2002 Nov;8(11):1227-34. doi: 10.1038/nm1102-1227. No abstract available. PMID 12411949
- [Background] Davi G, Patrono C. Platelet activation and atherothrombosis. N Engl J Med. 2007 Dec 13;357(24):2482-94. doi: 10.1056/NEJMra071014. No abstract available. PMID 18077812
- [Background] O'Kennedy N, Crosbie L, van Lieshout M, Broom JI, Webb DJ, Duttaroy AK. Effects of antiplatelet components of tomato extract on platelet function in vitro and ex vivo: a time-course cannulation study in healthy humans. Am J Clin Nutr. 2006 Sep;84(3):570-9. doi: 10.1093/ajcn/84.3.570. PMID 16960171
- [Background] Fuentes E, Forero-Doria O, Carrasco G, Marican A, Santos LS, Alarcon M, Palomo I. Effect of tomato industrial processing on phenolic profile and antiplatelet activity. Molecules. 2013 Sep 17;18(9):11526-36. doi: 10.3390/molecules180911526. PMID 24048285
- [Background] Fuentes E, Pereira J, Alarcon M, Valenzuela C, Perez P, Astudillo L, Palomo I. Protective Mechanisms of S. lycopersicum Aqueous Fraction (Nucleosides and Flavonoids) on Platelet Activation and Thrombus Formation: In Vitro, Ex Vivo and In Vivo Studies. Evid Based Complement Alternat Med. 2013;2013:609714. doi: 10.1155/2013/609714. Epub 2013 Sep 16. PMID 24159349
- [Background] Rodriguez-Azua R, Treuer A, Moore-Carrasco R, Cortacans D, Gutierrez M, Astudillo L, Fuentes E, Palomo I. Effect of tomato industrial processing (different hybrids, paste, and pomace) on inhibition of platelet function in vitro, ex vivo, and in vivo. J Med Food. 2014 Apr;17(4):505-11. doi: 10.1089/jmf.2012.0243. Epub 2013 Dec 10. PMID 24325459

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02986165/Prot_SAP_000.pdf